CLINICAL TRIAL: NCT00411827
Title: Goblet Cell Response and Dry Eye Symptoms After PRK and LASIK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Collaborators: Schepens Eye Research Institute (Other); State University of New York College of Optometry (Other)
Responsible Party: Principal Investigator, Samantha B. Rodgers, Assistant Director, Warfighter Refractive Eye Surgery Program and Research Center at FT Belvoir, Fort Belvoir Community Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WRAMC WU#06-23014
Record Dates: First submitted 2006-12-13; First posted 2006-12-15 (Estimated); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Keratoconjunctivitis Sicca
Keywords: Cytology; Keratomileusis, Laser In Situ; Keratectomy, Photorefractive, Excimer Laser
MeSH Terms: conditions — Keratoconjunctivitis Sicca | interventions — Postoperative Period; Keratomileusis, Laser In Situ

ARMS (2):
- 1 (Active Comparator): PRK
  Interventions: Procedure: PRK with conjunctival impression cytology before and after surgery
- 2 (Active Comparator): LASIK
  Interventions: Procedure: LASIK with conjunctival impression cytology before and after surgery

INTERVENTIONS:
Procedure: PRK with conjunctival impression cytology before and after surgery
  Arms: 1
Procedure: LASIK with conjunctival impression cytology before and after surgery — LASIK with conjunctival impression cytology before and after surgery
  Arms: 2

SUMMARY:
Purpose: To develop a screening metric by examining both the characteristics of the preoperative tear film and the intracellular signaling pathways of conjunctival goblet cells in order to determine if there are certain characteristics which might predict those patients who will experience serious dry eye symptoms and complications after refractive surgery.

Research Design: This study is a twelve-month prospective non-randomized investigation.

Methodology: In conjunction with psychometric questionnaires and various measures of tear film quality (e.g. Schirmer's test, tear break up time, etc), impression cytology will be used to assess the intracellular signaling pathways of conjunctival goblet cells and to determine if alterations in this pathway exist. Alterations in this pathway would result in a reduced response by the mucin secreting conjunctival goblet cells thereby promoting the development of dry eye after refractive surgery.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be recruited from those active duty soldiers that have requested refractive surgery. Subjects must be eligible for medical care at WRAMC.

1. Male or female, of any race, and at least 21 years old and not older than 40 years old at the time of the pre-operative examination, and have signed an informed consent. The lower age limit of 21 years is intended to ensure documentation of refractive stability and is the minimal age required by the FDA for informed consent for LASIK surgery.
2. Manifest refractive spherical equivalent (MSE) of up to 10.00 diopters at the spectacle plane with refractive cylinder up to 3.00 D.
3. Best spectacle corrected visual acuity of 20/20 or better in both eyes.
4. Patients who are willing to fill out dry eye questionnaires.
5. Demonstrated refractive stability, confirmed by clinical records. Neither the spherical nor the cylindrical portion of the refraction may have changed more than 0.50D during the 12- month period immediately preceding the baseline examination, as confirmed by clinical records.
6. All patients must be willing to return to the WRAMC Center for Refractive Surgery for follow up visits on Day1, Day 3, Day 7, and 1, 3, 6, and 12 months after their surgery.
7. Located in the greater Washington DC area for a 14-month period.
8. Consent of the subject's command (active duty) to participate in the study.
9. Access to transportation to meet follow-up requirements.

Exclusion Criteria:

1. Previous surgery or trauma to the study eye.
2. Dry eye as reflected by Schirmer's test with anesthesia of 0, subjective complaints or symptoms of dry eye, findings during the slit lamp exam that would be consistent with dry eye (e.g. superficial punctuate keratitis).
3. Female subjects who are pregnant, breast-feeding or intend to become pregnant during the study. This is a standard of care exclusion for refractive surgery at the Walter Reed Refractive Surgery Center because of the medications that are routinely given as part of the procedures. Standard of care analgesia consists of medications (e.g. narcotics) labeled as Pregnancy Category "C" by the FDA. Teratogenic effects are not known, however, physical dependence in the neonate may occur if the mother is given narcotics. Female subjects will be given a urine pregnancy test prior to participating in the study to rule out pregnancy.
4. Concurrent topical or systemic medications that may impair healing, including corticosteroids, antimetabolites, isotretinoin (Accutane), amiodarone hydrochloride (Cordarone) and/or sumatriptan (Imitrex).
5. Medical condition(s), which, in the judgment of the investigator, may impair healing, including but not limited to: collagen vascular disease, autoimmune disease, immunodeficiency diseases, and ocular herpes zoster or simplex.
6. Active ophthalmic disease, neovascularization of the cornea within 1mm of the intended ablation zone, or clinically significant lens opacity.
7. Evidence of glaucoma or an intraocular pressure greater than 22 mm Hg at baseline.
8. Evidence of keratoconus, corneal irregularity, or abnormal videokeratography in either eye.
9. History of recurrent erosions or epithelial basement dystrophy.
10. Patients with known sensitivity or inappropriate responsiveness to any of the medications used in the post-operative course.
11. Any physical or mental impairment that would preclude participation in any of the examinations.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 146 (Estimated)
Dates: Start 2008-01; Primary Completion 2011-02 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Dry eye | one year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Stutzman, MD, Principal Investigator — WRNMMC
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States